CLINICAL TRIAL: NCT04526340
Title: Food and Salt Handling in Diuresis: Research on Effects and Mechanisms of Food and Nutrients in Urine Output and Composition
Brief Title: Food and Salt Handling in Diuresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EC 2019/0710
Record Dates: First submitted 2020-08-12; First posted 2020-08-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nocturia; Polyuria
MeSH Terms: conditions — Nocturia; Polyuria | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutrient day (Experimental): on the nutrient day the subjects will take the testing food/nutrient capsules with 500 ml water
  Interventions: Diagnostic Test: Blood sample; Diagnostic Test: Bio-impedance measurement (BIA); Dietary Supplement: Ingestion of testing nutrient/food capsules; Diagnostic Test: Urine sample
- Control day (Placebo Comparator): on the control day the subjects will take 500 ml water without nutrient/food capsules
  Interventions: Diagnostic Test: Blood sample; Diagnostic Test: Bio-impedance measurement (BIA); Diagnostic Test: Urine sample

INTERVENTIONS:
Diagnostic Test: Blood sample — 2 Blood samples at the beginning and end of the test to analyze; Haptoglobin phenotyping, Haptoglobin concemtration (μmol/l) (serum), Sodium (mmol/l) (serum), Osmolality (mOsm/kg) (serum), Urea (g/l) (serum), Creatinine (g/dl) (serum), Potassium (mmol/l) (serum).
Diagnostic Test: Bio-impedance measurement (BIA) — for every 30 minutes for 4 hours
Dietary Supplement: Ingestion of testing nutrient/food capsules — The subjects will be tested in fasted and sober state in the morning. No food/drink 6 hours prior to the test. The subjects will be asked to take 2 different dosages of testing nutrient along with 500ml of water and only water for the control, on 3 different test days. The testing nutrients will be prepared in 1g capsules.
  Arms: Nutrient day
Diagnostic Test: Urine sample — 3 Urine samples at the beginning, after 2 hrs and at the end of the test to analyze: Total voided volume, Osmolality (mOsm/kg), Creatinine (g/dl), Sodium (mmol/l), Potassium (mmol/l), Urea (g/l)

SUMMARY:
Understanding the impact of food/nutrients on body fluid metabolism is important for improving diagnosis and treatment of nocturia, polyuria in relation to lifestyle interventions. This study on "Food and Salt Handling in Diuresis" examines the role of certain food and nutrients in diuresis. The study design is to investigate the possible acute effects and mechanisms of selected food (which are known to be diuretic) and nutrients (e.g. salt) in diuresis in healthy individuals. The study will provide insights into the management of nocturia, nocturnal polyuria or oedema which are common clinical sign in a wide range of disorders as cardiovascular, renal and metabolic disorders.

During the study the volunteers will be asked to ingest a certain dosage of a food/nutrient in capsules along with a defined amount of water (500 ml). 2 Blood and 3 urine samples will be collected at different time points to measure the urine output and urine composition derived by the ingestion of the particular food item. Renal Function Profiling is used as an easy and cheap tool to understand the mechanism of action behind the observed effect in diuresis. Renal function profiles distinguish the osmotic form water diuresis from a change in filtration.

Bio-electrical impedance analysis (BIA) is also used to evaluate oedema and fluid volumes in body tissues. BIA is a non-invasive technique based on Ohm's law whereby the resistance of a tissue against an electric current is inversely proportional to the water content and directly proportional to the length of the tissue. For the BIA measurement, a device is used in which 8 tactile electrodes are placed: 2 in contact with the thumb and middle finger of each hand, and 2 in contact with the inside and outside of each foot. Before the start of the measurements, the length and body weight are measured. The resistance of the arms, torso and legs is measured at different frequencies.

DETAILED DESCRIPTION:
Research design: Prospective intervention study to investigate the impact of food/nutrients on urine production and fluid distribution in the body.

Study sample: The sample size was calculated for a power of 80% and for control vs. treatment using a paired-sample t-test at the 5% significance level. Thus 30 young healthy volunteers for each food group (total 300 subjects for 10 food/nutrients groups as; leek, asparagus, onion, garlic, cranberry, barley, parsley, cardamom, coffee and salt) with no acute or chronic disease, no use of medication (except contraception), not being pregnant or menstruating at the time of the study, no any food allergies and age between 20-35 years with BMI 18.5-25 kg/m2 will be included. Volunteers with an implanted electronic device (e.g. Pacemaker) will not be included.

Methodology: The subjects will be tested in fasted and sober state in the morning. No food/drink 6hrs prior to the test. The subjects will be asked to take 2 different dosages of testing nutrient and along with 500ml of water and only 500ml water for the control, on 3 different test days. Nutrients will prepared in 1g capsules. The test will last for 4 hrs after taking of the capsules.

Analyses: 3-Days food diary: Once only. For salt, caffeine and energy intake Anthropometric measurements: at the beginning of each test day 2 Blood samples at the beginning and end of the test: Haptoglobin phenotyping (serum), Haptoglobin concentration (μmol/l) (serum), Sodium (mmol/l) (serum), Osmolality (mOsm/kg) (serum), Urea (g/l) (serum), Creatinine (g/dl) (serum) 3 Urine samples at the beginning, after 2 hrs and at the end of the test: Total voided volume, Osmolality (mOsm/kg), Creatinine (g/dl), Sodium (mmol/l), Potassium (mmol/l), Urea (g/l) Bio-impedance measurement (BIA): for every 30 min for 4 hours

Sample analysis and storage: Half of the urine samples and blood samples are sent immediately after collection to the university hospital Gent clinical laboratory. The other half of the samples will be stored for a certain time in a freezer at -80 °C and will be processed and examined for a second time. The other urine samples and blood samples that are not used for the research are stored as a bio-bank.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male/female
* Age between 20-35 years
* No use of medication (except contraception)
* Have no health issues
* Not being pregnant or menstruating at the time of the study
* BMI 18.5 -25 kg / m2
* No food allergies

Exclusion Criteria:

* Volunteers with an implanted electronic device (e.g. Pacemaker)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in urine volume (production) after ingestion of nutrient/food capsules | 4 hours
  the aim of this outcome is to check the effect on urine production after taking the capsules
Change in urine composition after ingestion of nutrient/food capsules | 4 hours
  the aim of this outcome is to check the effect on urine composition after taking the capsules
Change in serum composition after ingestion of nutrient/food capsules | 4 hours
  this aims to evaluate the effect in serum composition after taking the pills

SECONDARY OUTCOMES:
Change in body water distribution after ingestion of nutrients/food capsules | 4 hours
  using the bio-impedance measurement, the water distribution of the body over 4 hours is tested

CONTACTS AND LOCATIONS:
Overall Officials: Karel Everaert, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Department of Urology, Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No